CLINICAL TRIAL: NCT00101907
Title: An Open-Label, Dose-Finding Study to Evaluate the Safety of AMG 706 Plus Panitumumab Plus Gemcitabine-Cisplatin in the Treatment of Subjects With Advanced Cancer
Brief Title: Safety of AMG 706 Plus Panitumumab Plus Gemcitabine-Cisplatin in the Treatment of Patients With Advanced Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study terminated per recommendation of Data Review Team
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20040206
Record Dates: First submitted 2005-01-18; First posted 2005-01-19 (Estimated); Results first posted 2014-03-20 (Estimated); Last update posted 2014-03-20 (Estimated); Status verified 2014-02

CONDITIONS: Lung Cancer; Pancreatic Cancer; Esophageal Cancer
Keywords: Advanced Cancer; AMG 706; Panitumumab; Gemcitabine-Cisplatin
MeSH Terms: conditions — Lung Neoplasms; Pancreatic Neoplasms; Esophageal Neoplasms | interventions — motesanib diphosphate; Panitumumab; Gemcitabine; Cisplatin

ARMS (6):
- Panitumumab + Gem/Cis (Experimental): Panitumumab 9 mg/kg intravenously on Day 1 + gemcitabine (gem) 1250 mg/m^2 on Day 1 and Day 8, and cisplatin (cis) 75 mg/m^2 on Day 1 of each 3-week cycle.
  Interventions: Biological: Panitumumab; Drug: Gemcitabine; Drug: Cisplatin
- 50 mg QD AMG 706 + panitumumab + Gem/Cis (Experimental): AMG 706 50 mg administered orally once daily (QD) + panitumumab 9 mg/kg intravenously on Day 1 + gemcitabine (gem) 1250 mg/m^2 on Day 1 and Day 8, and cisplatin (cis) 75 mg/m^2 on Day 1 of each 3-week cycle.
  Interventions: Drug: AMG 706; Biological: Panitumumab; Drug: Gemcitabine; Drug: Cisplatin
- 75 mg QD AMG 706 + panitumumab + Gem/Cis (Experimental): AMG 706 75 mg administered orally once daily (QD) + panitumumab 9 mg/kg intravenously on Day 1 + gemcitabine (gem) 1250 mg/m^2 on Day 1 and Day 8, and cisplatin (cis) 75 mg/m^2 on Day 1 of each 3-week cycle.
  Interventions: Drug: AMG 706; Biological: Panitumumab; Drug: Gemcitabine; Drug: Cisplatin
- 100 mg QD AMG 706 + panitumumab + Gem/Cis (Experimental): AMG 706 100 mg administered orally once daily (QD) + panitumumab 9 mg/kg intravenously on Day 1 + gemcitabine (gem) 1250 mg/m^2 on Day 1 and Day 8, and cisplatin (cis) 75 mg/m^2 on Day 1 of each 3-week cycle.
  Interventions: Drug: AMG 706; Biological: Panitumumab; Drug: Gemcitabine; Drug: Cisplatin
- 125 mg QD AMG 706 + panitumumab + Gem/Cis (Experimental): AMG 706 125 mg administered orally once daily (QD) + panitumumab 9 mg/kg intravenously on Day 1 + gemcitabine (gem) 1250 mg/m^2 on Day 1 and Day 8, and cisplatin (cis) 75 mg/m^2 on Day 1 of each 3-week cycle.
  Interventions: Drug: AMG 706; Biological: Panitumumab; Drug: Gemcitabine; Drug: Cisplatin
- 75 mg BID AMG 706 + panitumumab + Gem/Cis (Experimental): AMG 706 75 mg administered orally twice daily (BID) + panitumumab 9 mg/kg intravenously on Day 1 + gemcitabine (gem) 1250 mg/m^2 on Day 1 and Day 8, and cisplatin (cis) 75 mg/m^2 on Day 1 of each 3-week cycle.
  Interventions: Drug: AMG 706; Biological: Panitumumab; Drug: Gemcitabine; Drug: Cisplatin

INTERVENTIONS:
Drug: AMG 706 — AMG 706 will be provided as 25-mg and 100-mg tablets and will be continuously self-administered orally once or twice daily based on cohort assignment starting on day 1 of Cycle 1.
  Arms: 100 mg QD AMG 706 + panitumumab + Gem/Cis; 125 mg QD AMG 706 + panitumumab + Gem/Cis; 50 mg QD AMG 706 + panitumumab + Gem/Cis; 75 mg BID AMG 706 + panitumumab + Gem/Cis; 75 mg QD AMG 706 + panitumumab + Gem/Cis
Biological: Panitumumab — Panitumumab will be administered by intravenous (IV) infusion at a dose of 9 mg/kg on Day 1 of each 3-week cycle.
  Other Names: Vectibix
Drug: Gemcitabine — Gemcitabine will be administered intravenously on Day 1 and Day 8 of each 21-day cycle at a dose of 1250 mg/m^2.
  Other Names: Gemzar
Drug: Cisplatin — Cisplatin will be administered intravenously on Day 1 of each 3-week cycle at a dose of 75 mg/m^2.
  Other Names: cisplatinum; cis-diamminedichloridoplatinum(II) (CDDP)

SUMMARY:
The purpose of this study is to characterize the safety and tolerability of AMG 706 plus panitumumab when administered with gemcitabine and cisplatin chemotherapy. This is a Phase 1b clinical study.

ELIGIBILITY:
For complete inclusion and exclusion, please refer to the investigator.

Inclusion Criteria:

* Competent to comprehend, sign, and date an Institutional Review Board (IRB) approved informed consent form
* Subjects with advanced cancer in whom the gemcitabine and cisplatin chemotherapy regimen is clinically indicated
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Adequate hematological function
* Adequate renal function
* Adequate hepatic function
* Life expectancy of greater than or equal to 3 months as documented by the investigator

Exclusion Criteria:

* More than 1 prior chemotherapy regimen
* History of venous thrombosis
* Myocardial infarction, cerebrovascular accident, transient ischemic attack, percutaneous transluminal coronary angioplasty/stent, or unstable angina within 1 year before study enrollment
* History of interstitial pneumonitis or pulmonary fibrosis or evidence of interstitial pneumonitis or pulmonary fibrosis on screening chest computed tomograph (CT) scan
* Average systolic blood pressure of greater than 145 mm Hg or average diastolic blood pressure of greater than 85 mm Hg
* Radiotherapy within 28 days of study enrollment or within 14 days of study enrollment for peripheral lesions
* Prior AMG 706, panitumumab, or another anti-EGFr monoclonal antibody (mAb) (e.g., cetuximab [Erbitux®] or EMD 72000)
* Systemic chemotherapy within 28 days before study enrollment
* Major surgery within 28 days or minor surgery within 14 days of study enrollment
* Central nervous system metastases (Exception: subjects with treated asymptomatic central nervous system metastases, those who have been clinically stable in the judgment of the investigator and off steroids for at least 30 days before the study enrollment are eligible)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2004-12; Primary Completion 2007-06 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Background] Burris H, Stephenson J, Otterson GA, Stein M, McGreivy J, Sun YN, Ingram M, Ye Y, Schwartzberg LS. Safety and pharmacokinetics of motesanib in combination with panitumumab and gemcitabine-Cisplatin in patients with advanced cancer. J Oncol. 2011;2011:853931. doi: 10.1155/2011/853931. Epub 2011 Apr 14. PMID 21559248
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 2 December 2004 through 7 March 2007. This study was designed with two parts. However, Part 2 was not conducted due to safety issues found in Part 1. Thus Part 1 is referenced as the overall study here.
Groups:
- Panitumumab + Gem/Cis: Panitumumab 9 mg/kg intravenously (IV) on Day 1 + gemcitabine (gem) 1250 mg/m^2 IV on Day 1 and Day 8, and cisplatin (cis) 75 mg/m^2 IV on Day 1 of each 3-week cycle.
- 50 mg QD AMG 706 + Panitumumab + Gem/Cis: AMG 706 50 mg administered orally once daily (QD) + panitumumab 9 mg/kg intravenously on Day 1 + gemcitabine 1250 mg/m^2 on Day 1 and Day 8, and cisplatin 75 mg/m^2 on Day 1 of each 3-week cycle.
- 75 mg QD AMG 706 + Panitumumab + Gem/Cis: AMG 706 75 mg administered orally once daily (QD) + panitumumab 9 mg/kg on Day 1 + gemcitabine 1250 mg/m^2 on Day 1 and Day 8, and cisplatin 75 mg/m^2 on Day 1 of each 3-week cycle.
- 100 mg QD AMG 706 + Panitumumab + Gem/Cis: AMG 706 100 mg administered orally once daily (QD) + panitumumab 9 mg/kg on Day 1 + gemcitabine 1250 mg/m^2 on Day 1 and Day 8, and cisplatin 75 mg/m^2 on Day 1 of each 3-week cycle.
- 125 mg QD AMG 706 + Panitumumab + Gem/Cis: AMG 706 125 mg administered orally once daily (QD) + panitumumab 9 mg/kg on Day 1 + gemcitabine 1250 mg/m^2 on Day 1 and Day 8, and cisplatin 75 mg/m^2 on Day 1 of each 3-week cycle.
- 75 mg BID AMG 706 + Panitumumab + Gem/Cis: AMG 706 75 mg administered orally twice daily (BID) + panitumumab 9 mg/kg on Day 1 + gemcitabine 1250 mg/m^2 on Day 1 and Day 8, and cisplatin 75 mg/m^2 on Day 1 of each 3-week cycle.
Period: Overall Study
Arm/Group | Panitumumab + Gem/Cis | 50 mg QD AMG 706 + Panitumumab + Gem/Cis | 75 mg QD AMG 706 + Panitumumab + Gem/Cis | 100 mg QD AMG 706 + Panitumumab + Gem/Cis | 125 mg QD AMG 706 + Panitumumab + Gem/Cis | 75 mg BID AMG 706 + Panitumumab + Gem/Cis
Started | 8 | 8 | 6 | 6 | 11 | 2
Completed | 6 | 7 | 5 | 5 | 6 | 2
Not Completed | 2 | 1 | 1 | 1 | 5 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 1 | 0 | 0 | 3 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Panitumumab + Gem/Cis: Panitumumab 9 mg/kg on Day 1 + gemcitabine (gem) 1250 mg/m^2 on Day 1 and Day 8, and cisplatin (cis) 75 mg/m^2 on Day 1 of each 3-week cycle.
- 50 mg QD AMG 706 + Panitumumab + Gem/Cis: AMG 706 50 mg administered orally once daily (QD) + panitumumab 9 mg/kg on Day 1 + gemcitabine 1250 mg/m^2 on Day 1 and Day 8, and cisplatin 75 mg/m^2 on Day 1 of each 3-week cycle.
- 100 mg QD AMG 706 + Panitumumab + Gem/Cis: AMG 706 100 mg administered orally once daily + panitumumab 9 mg/kg on Day 1 + gemcitabine 1250 mg/m^2 on Day 1 and Day 8, and cisplatin 75 mg/m^2 on Day 1 of each 3-week cycle.
- 125 mg QD AMG 706 + Panitumumab + Gem/Cis: AMG 706 125 mg administered orally once daily + panitumumab 9 mg/kg on Day 1 + gemcitabine 1250 mg/m^2 on Day 1 and Day 8, and cisplatin 75 mg/m^2 on Day 1 of each 3-week cycle.
- Total: Total of all reporting groups
Arm/Group | Panitumumab + Gem/Cis | 50 mg QD AMG 706 + Panitumumab + Gem/Cis | 75 mg QD AMG 706 + Panitumumab + Gem/Cis | 100 mg QD AMG 706 + Panitumumab + Gem/Cis | 125 mg QD AMG 706 + Panitumumab + Gem/Cis | 75 mg BID AMG 706 + Panitumumab + Gem/Cis | Total
Number analyzed (Participants) | 8 | 8 | 6 | 6 | 11 | 2 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.5 (12.4) | 60.4 (13.8) | 56.0 (13.3) | 51.5 (13.5) | 61.1 (8.3) | 65.0 (17.0) | 57.9 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 2 | 4 | 5 | 0 | 18
  Male | 4 | 5 | 4 | 2 | 6 | 2 | 23
Race/Ethnicity, Customized [Number; unit: Participants]
  Black or African American | 1 | 1 | 2 | 0 | 0 | 0 | 4
  Hispanic or Latino | 1 | 0 | 0 | 0 | 0 | 0 | 1
  White or Caucasian | 6 | 7 | 4 | 6 | 11 | 2 | 36

OUTCOME MEASURES:

1. Secondary Outcome: Number of Participants With an Objective Tumor Response
Description: The number of participants with a confirmed objective tumor response, defined as a complete response (CR) or partial response (PR) throughout based on modified Response Evaluation Criteria in Solid Tumors (RECIST) criteria. Any CR or PR was to be confirmed 4 to 6 weeks after the initial CR or PR.
Time Frame: From enrollment until date of last follow-up visit. The median follow-up time was 24 weeks, with a range of 3 to 73 weeks.
Population: Efficacy Analysis Set, defined as defined as patients who received at least 1 dose of AMG 706 for AMG 706 treatment groups and patients who received at least 1 dose of panitumumab for the panitumumab-only treatment group.
Measure: Number; unit: participants
Arm/Group | Panitumumab + Gem/Cis | 50 mg QD AMG 706 + Panitumumab + Gem/Cis | 75 mg QD AMG 706 + Panitumumab + Gem/Cis | 100 mg QD AMG 706 + Panitumumab + Gem/Cis | 125 mg QD AMG 706 + Panitumumab + Gem/Cis | 75 mg BID AMG 706 + Panitumumab + Gem/Cis
Number analyzed (Participants) | 8 | 8 | 6 | 6 | 11 | 2
participants | 2 | 0 | 1 | 4 | 2 | 1

2. Secondary Outcome: Tmax
Description: Time after dosing when maximum plasma concentration was observed for AMG 706
Time Frame: Day 1, pre-dose and at 1, 3, 6,12 (BID cohort only) and 24 hours post-dose.
Population: The Pharmacokinetic (PK) Analysis Set consists of patients who had dosing and PK sampling times recorded on the day of PK sample collection and no significant protocol deviations that impacted the quality of the PK data (for example, sample processing errors and/or inaccurate dosing on the day of the PK sampling).
Measure: Median (Full Range); unit: hours
Arm/Group | 50 mg QD AMG 706 + Panitumumab + Gem/Cis | 75 mg QD AMG 706 + Panitumumab + Gem/Cis | 100 mg QD AMG 706 + Panitumumab + Gem/Cis | 125 mg QD AMG 706 + Panitumumab + Gem/Cis | 75 mg BID AMG 706 + Panitumumab + Gem/Cis
Number analyzed (Participants) | 8 | 6 | 4 | 11 | 2
hours | 1.00 [1.00 to 3.00] | 1.00 [1.00 to 3.00] | 1.38 [1.00 to 3.00] | 1.00 [1.00 to 3.00] | 1.00 [1.00 to 1.00]

3. Secondary Outcome: Cmax
Description: The maximum observed plasma concentration after AMG 706 dosing
Time Frame: Day 1, pre-dose and at 1, 3, 6,12 (BID cohort only) and 24 hours post-dose.
Population: PK analysis set.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 50 mg QD AMG 706 + Panitumumab + Gem/Cis | 75 mg QD AMG 706 + Panitumumab + Gem/Cis | 100 mg QD AMG 706 + Panitumumab + Gem/Cis | 125 mg QD AMG 706 + Panitumumab + Gem/Cis | 75 mg BID AMG 706 + Panitumumab + Gem/Cis
Number analyzed (Participants) | 8 | 6 | 4 | 11 | 2
ng/mL | 152 (78) | 186 (92) | 278 (90) | 458 (208) | 268 (NA) — Standard deviation could not be calculated due to sample size of 2.

4. Secondary Outcome: AUC0-24
Description: Area under the plasma concentration-time curve from time 0 to 24 hours postdose (AUC0-24) with AMG 706. AUC0-24 was estimated using the linear/log trapezoidal method. For the BID cohort, AUC0 24 was estimated as 2 times the AUC from time 0 to 12 hours post the first daily dose (AUC0-12) using the linear/log trapezoidal method.
Time Frame: Day 1, pre-dose and at 1, 3, 6,12 (BID cohort only) and 24 hours post-dose.
Population: PK Analysis set; Patients with elevated AMG 706 concentrations at 24 hours were excluded from the AUC summary statistics calculations.
Measure: Mean (Standard Deviation); unit: μg*hr/mL
Arm/Group | 50 mg QD AMG 706 + Panitumumab + Gem/Cis | 75 mg QD AMG 706 + Panitumumab + Gem/Cis | 100 mg QD AMG 706 + Panitumumab + Gem/Cis | 125 mg QD AMG 706 + Panitumumab + Gem/Cis | 75 mg BID AMG 706 + Panitumumab + Gem/Cis
Number analyzed (Participants) | 7 | 4 | 2 | 11 | 2
μg*hr/mL | 1.03 (0.50) | 1.31 (0.51) | 2.38 (NA) — Standard deviation could not be calculated due to sample size of 2. | 2.82 (1.02) | 2.54 (NA) — Standard deviation could not be calculated due to sample size of 2.

5. Secondary Outcome: AUC0-inf
Description: Area under the concentration-time curve from time 0 to infinite time (AUC0-inf) postdose with AMG 706. AUC0-inf was estimated using the linear/log trapezoidal method. AUC0-inf was not calculated for the BID cohort.
Time Frame: Day 1, pre-dose and at 1, 3, 6,12 (BID cohort only) and 24 hours post-dose.
Population: PK analysis set. Patients with elevated AMG 706 concentrations at 24 hours were excluded from the AUC summary statistics calculations.
Measure: Mean (Standard Deviation); unit: μg*hr/mL
Arm/Group | 50 mg QD AMG 706 + Panitumumab + Gem/Cis | 75 mg QD AMG 706 + Panitumumab + Gem/Cis | 100 mg QD AMG 706 + Panitumumab + Gem/Cis | 125 mg QD AMG 706 + Panitumumab + Gem/Cis | 75 mg BID AMG 706 + Panitumumab + Gem/Cis
Number analyzed (Participants) | 7 | 3 | 2 | 9 | 0
μg*hr/mL | 1.12 (0.52) | 1.64 (0.48) | 2.59 (NA) — Standard deviation not calculated due to sample size of 2. | 3.05 (1.34) |

6. Primary Outcome: Participant Incidence of Adverse Events
Description: The number of participants who experienced at least one treatment-emergent adverse event. Additional details regarding specfic adverse events are provided in the Adverse Event section of this posting.
Time Frame: From the first dose of any study treatment until 30 days after the last dose of study treatment, up to a maximum of 509 days.
Population: Safety Analysis Set, composed of all participants in the AMG 706 treatment groups who received at least one dose of AMG 706 and all participants in the panitumumab-only treatment group who received at least one dose of panitumumab.
Measure: Number; unit: Participants
Groups:
- 100 mg QD AMG 706 + Panitumumab + Gem/Cis: AMG 706 100 mg administered orally once daily (QD) + panitumumab 9 mg/kg intravenously on Day 1 + gemcitabine 1250 mg/m^2 on Day 1 and Day 8, and cisplatin 75 mg/m^2 on Day 1 of each 3-week cycle.
Arm/Group | Panitumumab + Gem/Cis | 50 mg QD AMG 706 + Panitumumab + Gem/Cis | 75 mg QD AMG 706 + Panitumumab + Gem/Cis | 100 mg QD AMG 706 + Panitumumab + Gem/Cis | 125 mg QD AMG 706 + Panitumumab + Gem/Cis | 75 mg BID AMG 706 + Panitumumab + Gem/Cis
Number analyzed (Participants) | 8 | 8 | 6 | 6 | 11 | 2
Participants | 8 | 8 | 6 | 6 | 11 | 2

ADVERSE EVENTS:
Time Frame: From the first dose of any study treatment until 30 days after the last dose of study treatment, up to a maximum of 509 days.
Description: The table of Other Adverse Events summarizes the most frequent non-serious occurrences of adverse events.
Groups:
- 125 mg QD AMG 706 + Panitumumab + Gem/CisEdit: AMG 706 125 mg administered orally once daily (QD) + panitumumab 9 mg/kg on Day 1 + gemcitabine 1250 mg/m^2 on Day 1 and Day 8, and cisplatin 75 mg/m^2 on Day 1 of each 3-week cycle.
- 75 mg BID AMG 706 + Panitumumab + Gem/CisEdit: AMG 706 75 mg administered orally twice daily (BID) + panitumumab 9 mg/kg on Day 1 + gemcitabine 1250 mg/m^2 on Day 1 and Day 8, and cisplatin 75 mg/m^2 on Day 1 of each 3-week cycle.
Arm/Group | Panitumumab + Gem/Cis | 50 mg QD AMG 706 + Panitumumab + Gem/Cis | 75 mg QD AMG 706 + Panitumumab + Gem/Cis | 100 mg QD AMG 706 + Panitumumab + Gem/Cis | 125 mg QD AMG 706 + Panitumumab + Gem/CisEdit | 75 mg BID AMG 706 + Panitumumab + Gem/CisEdit
Serious Adverse Events (participants affected / at risk) | 2/8 | 4/8 | 3/6 | 4/6 | 9/11 | 1/2
Other Adverse Events (participants affected / at risk) | 8/8 | 8/8 | 6/6 | 6/6 | 11/11 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Panitumumab + Gem/Cis (N=8) | 50 mg QD AMG 706 + Panitumumab + Gem/Cis (N=8) | 75 mg QD AMG 706 + Panitumumab + Gem/Cis (N=6) | 100 mg QD AMG 706 + Panitumumab + Gem/Cis (N=6) | 125 mg QD AMG 706 + Panitumumab + Gem/CisEdit (N=11) | 75 mg BID AMG 706 + Panitumumab + Gem/CisEdit (N=2)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 1 | 0 | 0 | 0 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
Anal fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Oesophageal perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 1 | 1 | 0 | 0
Sudden death (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Catheter related infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Narcotic intoxication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 3 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1 | 3 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Arterial thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 2 | 0 | 1 | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Panitumumab + Gem/Cis (N=8) | 50 mg QD AMG 706 + Panitumumab + Gem/Cis (N=8) | 75 mg QD AMG 706 + Panitumumab + Gem/Cis (N=6) | 100 mg QD AMG 706 + Panitumumab + Gem/Cis (N=6) | 125 mg QD AMG 706 + Panitumumab + Gem/CisEdit (N=11) | 75 mg BID AMG 706 + Panitumumab + Gem/CisEdit (N=2)
Anaemia (Blood and lymphatic system disorders) | 6 | 5 | 2 | 5 | 4 | 1
Haemorrhagic diathesis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypocoagulable state (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 4 | 5 | 4 | 5 | 3 | 0
Polycythaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 5 | 2 | 2 | 5 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 | 1 | 0
Cardiac tamponade (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cardiomegaly (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1 | 1 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Supraventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 1 | 0 | 0 | 0
Deafness (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 1
Ear congestion (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hearing impaired (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0
Middle ear effusion (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 2 | 1 | 1 | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0
Conjunctivitis (Eye disorders) | 0 | 1 | 0 | 0 | 1 | 0
Diplopia (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Erythema of eyelid (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Eye swelling (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Eyelid oedema (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Eyelids pruritus (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 1 | 1 | 1 | 0 | 0 | 0
Visual disturbance (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 5 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Chapped lips (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 3 | 3 | 3 | 3 | 6 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 4 | 4 | 9 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 2 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Eructation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1 | 1 | 2 | 3 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Gingival disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hyperchlorhydria (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Lip dry (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 6 | 6 | 5 | 6 | 10 | 1
Rectal discharge (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 1 | 2 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 4 | 4 | 3 | 4 | 6 | 0
Adverse drug reaction (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Application site rash (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Asthenia (General disorders) | 0 | 2 | 0 | 0 | 2 | 0
Catheter site discharge (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Catheter site erythema (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Catheter site pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Catheter site related reaction (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Crepitations (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cyst (General disorders) | 1 | 0 | 0 | 0 | 0 | 1
Early satiety (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Extravasation (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 5 | 7 | 3 | 4 | 10 | 2
Generalised oedema (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypothermia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Impaired healing (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Infusion site reaction (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Injection site bruising (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Injection site reaction (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Mucosal inflammation (General disorders) | 4 | 1 | 0 | 5 | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 1 | 0 | 0 | 0 | 0
Oedema (General disorders) | 0 | 1 | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 1 | 1 | 2 | 2 | 0 | 1
Pain (General disorders) | 1 | 1 | 1 | 1 | 2 | 0
Pyrexia (General disorders) | 1 | 1 | 1 | 1 | 0 | 0
Gallbladder disorder (Hepatobiliary disorders) | 0 | 0 | 1 | 1 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Adenoviral conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Candidiasis (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0
Catheter related infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 2 | 0 | 0
Conjunctivitis viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Infected sebaceous cyst (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Localised infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0
Nail bed infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 2 | 0
Onychomycosis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0
Oral fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0
Paronychia (Infections and infestations) | 3 | 0 | 0 | 1 | 2 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Rash pustular (Infections and infestations) | 0 | 1 | 0 | 1 | 2 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Tinea pedis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 1 | 3 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 2 | 1 | 0 | 0
Aspartate aminotransferase (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 1 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Blood magnesium decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Blood phosphorus decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Blood potassium decreased (Investigations) | 1 | 0 | 1 | 0 | 0 | 0
Breath sounds abnormal (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 1 | 0 | 0 | 2 | 0
International normalised ratio increased (Investigations) | 0 | 1 | 1 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 2 | 1 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Platelet count increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Prothrombin time ratio increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Weight decreased (Investigations) | 1 | 0 | 3 | 1 | 5 | 0
Anorexia (Metabolism and nutrition disorders) | 4 | 4 | 0 | 4 | 6 | 0
Appetite disorder (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 0 | 1 | 0 | 3 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypercreatininaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 4 | 6 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 3 | 3 | 3 | 6 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 2 | 3 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 3 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1 | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 2 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 2 | 2 | 3 | 2 | 0
Dysarthria (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 2 | 2 | 1 | 3 | 4 | 0
Facial palsy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 2 | 2 | 1 | 2 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 2 | 0 | 1 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 2 | 1 | 1 | 0
Sinus headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Abnormal dreams (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 1 | 3 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 2 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 4 | 0
Insomnia (Psychiatric disorders) | 0 | 3 | 2 | 2 | 4 | 0
Libido decreased (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Mood altered (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Sleep disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1 | 1 | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Breast tenderness (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 5 | 1 | 2 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2 | 2 | 4 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0 | 1 | 0
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 2 | 4 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 2 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 1 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 3 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 2 | 2 | 5 | 3 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 5 | 5 | 4 | 4 | 4 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 2 | 2 | 1 | 2 | 1
Erythema (Skin and subcutaneous tissue disorders) | 5 | 5 | 6 | 5 | 3 | 1
Exfoliative rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 2 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Increased tendency to bruise (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 2 | 5 | 5 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 6 | 5 | 2 | 4 | 3 | 2
Rash erythematous (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 3 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 2 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 1 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Central venous catheterisation (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 1 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hot flush (Vascular disorders) | 1 | 0 | 1 | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 3 | 4 | 2 | 5 | 1
Hypotension (Vascular disorders) | 0 | 1 | 1 | 1 | 0 | 0
Jugular vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Venous thrombosis limb (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results aftercompletion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.